CLINICAL TRIAL: NCT02217631
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics (Biomarkers) of BI 653048 BS H3PO4 Capsule Formulation Administered as Multiple Doses of 25 mg to 200 mg qd for 10 Days. A Randomised, Double-blind Within Dose Groups, Placebo-controlled, Multiple Rising Dose Trial With Open-label Active Comparator
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BI 653048 BS H3PO4 Capsule Multiple Rising Doses in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1262.2
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — BI 653048 BS H3PO4; Prednisolone

ARMS (4):
- BI 653048 BS H3PO4 (Experimental): dose escalation
  Interventions: Drug: BI 653048 BS H3PO4
- Prednisolone low dose (Active Comparator)
  Interventions: Drug: Prednisolone low dose
- Prednisolone high dose (Active Comparator)
  Interventions: Drug: Prednisolone high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 653048 BS H3PO4
  Arms: BI 653048 BS H3PO4
Drug: Prednisolone low dose
  Arms: Prednisolone low dose
Drug: Prednisolone high dose
  Arms: Prednisolone high dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objectives of the trial were to assess safety, tolerability, pharmacokinetics, and pharmacodynamics of multiple rising doses of BI 653048 BS H3PO4 compared with prednisolone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects based on a complete medical history, physical examination, vital signs (blood pressure and pulse rate), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 50 years
* Body mass index (BMI) of 18.5 to 29.9 kg/m2
* Signed and dated written informed consent in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any clinically relevant deviation from normal in the medical examination including blood pressure, pulse rate, and ECG
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy), psychiatric disorders, or neurological disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 h) within at least 1 month or less than 10 half-lives of the respective drug before first treatment with study drug or during trial
* Use of drugs which might reasonably influence the results of the trial or which prolong the QT/QTc interval within 10 days before first treatment with study drug or during trial
* Participation in another trial with an investigational drug within 30 days before first treatment with study drug or during trial
* Smoker (more than 10 cigarettes, 3 cigars, or 3 pipes per day)
* Inability to refrain from smoking beginning from 1 day before first treatment with study drug until discharge from the clinical unit
* Alcohol abuse (more than 60 grams per day)
* Drug abuse
* Blood donation of more than 100 mL within 4 weeks before first treatment with study drug or during trial
* Excessive physical activities within 1 week before first treatment with study drug or during trial
* Any laboratory value outside the reference range and of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of the QT/QTc interval (e.g. QTc intervals that are repeatedly longer than 450 ms)
* A history of additional risk factors for torsades de points (e.g. heart failure, hypokalaemia, or family history of Long QT syndrome

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to day 14
Number of patients with clinically significant findings in vital signs | up to 10 days after last drug administration
  blood pressure, pulse rate, body temperature, orthostatic test
Number of patients with clinically significant findings in ECG | up to 10 days after last drug administration
Number of patients with clinically significant findings in laboratory tests | up to 10 days after last drug administration
Assessment of tolerability by the investigator on a four-point scale | up to 10 days after last drug administration

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in plasma at different time points (Cmax) | up to day 13
time from dosing to maximum measured concentration of the analyte at different time points (tmax) | up to day 13
Area under the concentration-time curve of the analyte in the plasma over time interval from 0 to the last measurable time point of the dose at different time points (AUC0-tz) | up to day 13
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity at different time points (AUC0-∞) | up to day 13
Percentage of the AUC0-∞ that is obtained by extrapolation at different time points (%AUCtz-∞) | up to day 13
Terminal phase elimination rate constant at different time points (λz) | up to day 13
Mean residence time of the analyte in the body after oral administration at different time points (MRTpo) | up to day 13
Terminal phase elimination half life at different time points (t1/2) | up to day 13
Apparent clearance of the analyte in plasma following extravascular administration at steady state (CL/Fss) | up to day 13
Apparent volume of distribution during the terminal phase λz following an extravascular dose at steady state (Vz/Fss) | up to day 13
Minimum plasma concentration at steady state (Cmin,ss) | up to day 13
Dose-normalized Cmax at steady state (Cmax/Dss) | up to day 13
Dose-normalised AUC0-∞ at steady state (AUC0-∞/Dss) | up to day 13
Accumulation index of the analyte when comparing AUCτ (RA,AUCτ) | up to day 13
Accumulation index of the analyte when comparing Cmax (RA,Cmax) | up to day 13
Linearity index (LI) | up to day 13
Amount of analyte excreted in urine unchanged from t1 to t2 interval at different time points (Aet1-t2) | up to day 11
Renal clearance of the unchanged analyte at different time points (CLr) | up to day 11
Area under the serum biomarker concentration-time curve after the Nth dose (AUECN) | up to day 13
Area under the baseline (before dose level) but above serum biomarker concentration-time curve after the Nth dose (AUECbelow_base) | up to day 13
Minimum measured serum concentration of the biomarkers after the Nth dose (Emin,N) | up to day 13
Maximum measured serum concentration of the biomarkers after the Nth dose (Emax,N) | up to day 13
Serum biomarker concentration after the (N-1)th dose but before the Nth dose (Epre,N) | up to day 13
Measured value of the biomarkers in biological matrix at the set time point after Nth dose (EN) | up to day 13
Oral glucose insulin sensitivity (OGIS) index | up to day 13
Homeostasis model assessment (HOMA) value | up to day 13

REFERENCES:
- [Derived] Harcken C, Scholl P, Nabozny G, Thomson D, Bianchi D. Clinical profile of the functionally selective glucocorticoid receptor agonist BI 653048 in healthy male subjects. Expert Opin Investig Drugs. 2019 May;28(5):489-496. doi: 10.1080/13543784.2019.1599859. Epub 2019 Apr 9. PMID 30908082